CLINICAL TRIAL: NCT01875679
Title: Surgical Coaching -Using Error Debriefing, Behavioral Modeling and Error Recognition to Enhance Surgical Skill
Brief Title: Comprehensive Surgical Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CSC2013
Record Dates: First submitted 2013-05-15; First posted 2013-06-12 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Surgical Technical Skill; Technical Errors in Surgery
Keywords: Surgical education; Deliberate practice; Debriefing; Behaviour modelling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional residency training (Active Comparator): This group will continue their regular surgical training without any specific intervention.
  Interventions: Other: Conventional Surgical Training
- Comprehensive Surgical Coaching (SCS) (Experimental): The participants will receive an analysis of the technical performance as observed on baseline recordings of the index procedure. Training needs will be identified and a personalized coaching concept will be designed. Coaching sessions will include video debriefing of the participant's performance (sample recordings will be submitted by the participant during the sessions) and video assisted behavioral modeling using examples of good and poor technical performance. Coaching will also target increasing awareness of weaknesses and potential pitfalls in surgical technical task execution (error recognition).
  Interventions: Other: Comprehensive Surgical Coaching

INTERVENTIONS:
Other: Comprehensive Surgical Coaching
  Arms: Comprehensive Surgical Coaching (SCS)
Other: Conventional Surgical Training — Surgical training as per participant's residency program
  Arms: Conventional residency training

SUMMARY:
Simulation in surgical skills training is widely accepted as a necessary step to improve surgical training outside the operating room. Simulation predominately focuses on teaching a specific task or procedure. Once this task is acquired ongoing optimization of technique is desirable. Commonly ongoing skills assessment occurs in the form of peer feedback throughout training rotations. This feedback is frequently subjective and of variable educational use. Identifying ongoing technical training needs and enabling personalized objective feedback represents an important training concept that has not yet been formally used in resident training.

The specific goal of this study is to prove the effect of a comprehensive surgical coaching (CSC) approach which combines concepts of behavior modeling training, task debriefing and error recognition to improve overall surgical technique without additional technical skills training.

DETAILED DESCRIPTION:
Design The study design is a randomized, controlled trial involving evaluation of a study and a conventionally trained group at pretest and posttest.

Participants The study and control groups will consist of senior surgical residents (PGY 3-5) and surgical fellows involved in minimally invasive surgery (MIS).

Inclusion: Since concurrent operative training in the operating room (OR) in the technique of MIS is a prerequisite for this study, only residents and fellows on rotations with a practice focus on MIS during the time period of the study will be eligible for participation.

Exclusion: Individuals with severe illnesses precluding performance in the OR will not be included.

Outcome measures: Surgical performance will be assessed using a global rating scale as well as through tabulation of observed intraoperative technical errors. Primary outcome measure is surgical skill level before and after targeted training.

ELIGIBILITY:
Inclusion Criteria:

* surgical residents and fellows on rotations with a practice focus on minimally invasive surgery during the time period of the study

Exclusion Criteria:

* individuals with severe illnesses precluding performance in the OR

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Surgical Technical Skill | After 8 weeks of participation
  Surgical skill measures as recorded on a procedure specific global rating scale, Objective Structured Assessment of Technical Skills (OSATS) and bariatric OSATS (BOSATS) scores and by tabulation of technical errors, Generic Error Rating Tool (GERT) observed during the index procedures.

SECONDARY OUTCOMES:
Learning curves | Throughout 8 weeks of participation
  Development of skill and reduction of errors will be assessed in relation to number of procedures performed to obtain learning curves for each study group.
  Surgical technical skill will be assessed by OSATS and BOSATS scales, errors will be recorded by GERT checklist

CONTACTS AND LOCATIONS:
Overall Officials: Teodor P Grantcharov, MD. PhD, Principal Investigator — St. Michael's Hospital (Toronto, Canada)
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada